CLINICAL TRIAL: NCT02353013
Title: Effect of Protein Intake on Preterm Infant Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Courtney B. Atchley, DO, Assistant Professor of Pediatrics, University of Oklahoma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4885
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Premature; Infant, Light-for-dates
Keywords: protein intake; body composition
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Protein Group (Active Comparator): For infants in this group, the target protein-energy ratio (PER) will be ~3 g/100 kcal. This will be achieved by providing standard fortification by adding a commercially available human milk fortifier to human milk or by providing a preterm formula.
  Interventions: Dietary Supplement: Standard fortification
- Enhanced Protein Group (Experimental): For infants in this group, the target protein-energy ratio (PER) will be ~4 g/100 kcal. This will be achieved by providing standard fortification by adding a commercially available human milk fortifier to human milk or by providing a preterm formula. In addition, liquid protein will be added to provide protein supplementation and increase the PER.
  Interventions: Dietary Supplement: Protein supplementation; Dietary Supplement: Standard fortification

INTERVENTIONS:
Dietary Supplement: Protein supplementation — Standard fortification of human milk may not have enough protein for optimal growth of premature infants. The investigators will add extra protein to this group to increase the protein consumed.
  Arms: Enhanced Protein Group
Dietary Supplement: Standard fortification — Standard fortification of human milk involves adding a commercially available human milk fortifier to human milk in order to increase several nutrients.

SUMMARY:
The investigators will compare weight gain based on fat accretion and change in body composition in preterm infants receiving different amounts of enteral protein.

DETAILED DESCRIPTION:
American Academy of Pediatrics guidelines define the growth rate of preterm, underweight babies as adequate if it matches the age-equivalent weight gains typical of term infants, approximately 10-15 grams per kg per day. Unfortunately, many pre-terms, especially very low birth weight ones, do not achieve this rate, resulting in neurodevelopmental deficits and low discharge weights. Typical feeding regimens, designed to increase weight gain, however, have been shown to increase the rate of fat accretion and increase the risk of obesity and metabolic disorders, such as insulin resistance and type 2 diabetes, later in life. Research has shown that higher protein diets can reduce the accretion of body fat in older, normal weight infants but this has not been systematically tested in low birth weight pre-terms. The current study will compare weight gain based on fat accretion and change in body composition in preterm infants receiving higher (4g/100 kcal) versus lower (3 g/100 kcal) protein-energy ratio diets. The hypothesis tested in this study is: Increased protein intake will reduce the percentage of weight gain due to fat accretion in pre-term infants. The identification of an effective feeding regimen that would both allow pre-term infants to acquire age-equivalent growth rates similar to those of term infants while avoiding the excess accretion of body fat could significantly improve the long term health outcomes of this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants born less than 32 weeks EGA
* Growth that is appropriate for gestational age (AGA)
* Admitted to OU Children's NICU, inborn or outborn
* Receiving enteral feedings <100 mL/kg/day
* Hemodynamically stable

Exclusion Criteria:

* Severe congenital anomalies to include congenital heart disease, chromosomal anomalies, open neural tube defects, and/or intestinal anomalies precluding enteral feedings
* Growth restriction, growth that is small for gestational age (SGA) or large for gestational age (LGA)
* Inborn errors of metabolism
* History of necrotizing enterocolitis Bell stage III
* Cerebrospinal fluid indwelling shunt (affects body composition measurements)
* Expected death prior to 36 weeks EGA (the end of the study period)
* Inability to meet Pea Pod® requirements for the first measurement
* On vasopressor medications

Ages: 1 Minute to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2014-12; Primary Completion 2017-07 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Weight gain due to fat mass | 4 weeks

SECONDARY OUTCOMES:
Change in body weight | 4 weeks
Change in percent fat mass | 4 weeks
Change in length | 4 weeks
Change in head circumference | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Courtney B Atchley, DO, Principal Investigator — OUHSC
Locations (1):
- OUHSC Children's Hospital, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atchley CB, Cloud A, Thompson D, Blunt MH, Satnes KJ, Szyld E, Ernst KD. Enhanced Protein Diet for Preterm Infants: A Prospective, Randomized, Double-blind, Controlled Trial. J Pediatr Gastroenterol Nutr. 2019 Aug;69(2):218-223. doi: 10.1097/MPG.0000000000002376. PMID 31058772